CLINICAL TRIAL: NCT00008333
Title: Oral Vinorelbine For The Treatment Of Metastatic Non-Small Cell Lung Cancer In Patients More Than Or Equal To 65 Years Of Age: A Phase II Trial of Efficacy and Patients Perceived Preference for Oral Therapy
Brief Title: Vinorelbine in Treating Older Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0022; NCI-2012-02369 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068398 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-01-06; First posted 2004-02-03 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vinorelbine (Experimental): Patients receive oral vinorelbine on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and after 8 weeks of therapy. Patients are followed every 3 months for 5 years.
  Interventions: Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine taken by mouth in treating older patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in elderly patients with stage IIIB or IV non-small cell lung cancer treated with oral vinorelbine. II. Determine the time to progression in patients treated with this drug. III. Determine the toxicity of this drug in these patients. IV. Determine whether there is a perceived preference for this oral administration in these patients. V. Determine the quality of life of these patients when treated with this drug. VI. Assess individual variation in responses, pharmacokinetic parameters, and/or biological correlates in patients treated with this drug.

OUTLINE: Patients receive oral vinorelbine on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and after 8 weeks of therapy. Patients are followed every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIIB or IV non-small cell lung cancer Measurable disease At least 1 lesion that is 2.0 cm or more in longest diameter CNS metastases allowed if previously treated and clinically stable for at least 8 weeks prior to study No meningeal carcinomatosis Participation in translational research component of this study is mandatory

PATIENT CHARACTERISTICS: Age: 65 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Platelet count at least 100,000/mm3 Hemoglobin at least 10.0 g/dL Absolute neutrophil count at least 1,500/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2 times upper limit of normal Other: No dysphagia or inability to swallow capsules intact No peripheral neuropathy grade 2 or greater No other significant medical condition that would preclude study No active infection within the past 2 weeks No other malignancy within the past 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for this disease within the past 5 years Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No prior radiotherapy to more than 25% of bone marrow No prior radiotherapy to measurable lesion unless documented progression after therapy No concurrent radiotherapy, including palliative radiotherapy Surgery: At least 3 weeks since prior major surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2001-04; Primary Completion 2004-03 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
objective response rate | Up to 5 years

SECONDARY OUTCOMES:
Time to progression | Up to 5 years
Quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (13):
- United States (13):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Background] Huschka MM, Mandrekar SJ, Schaefer PL, Jett JR, Sloan JA. A pooled analysis of quality of life measures and adverse events data in north central cancer treatment group lung cancer clinical trials. Cancer. 2007 Feb 15;109(4):787-95. doi: 10.1002/cncr.22444. PMID 17211864
- [Background] Jatoi A, Hillman S, Stella P, Green E, Adjei A, Nair S, Perez E, Amin B, Schild SE, Castillo R, Jett JR; North Central Cancer Treatment Group. Should elderly non-small-cell lung cancer patients be offered elderly-specific trials? Results of a pooled analysis from the North Central Cancer Treatment Group. J Clin Oncol. 2005 Dec 20;23(36):9113-9. doi: 10.1200/JCO.2005.03.7465. PMID 16361618
- [Result] Kanard A, Jatoi A, Castillo R, Geyer S, Schulz TK, Fitch TR, Rowland KM, Nair S, Krook JE, Kugler JW. Oral vinorelbine for the treatment of metastatic non-small cell lung cancer in elderly patients: a phase II trial of efficacy and toxicity. Lung Cancer. 2004 Mar;43(3):345-53. doi: 10.1016/j.lungcan.2003.09.012. PMID 15165094